CLINICAL TRIAL: NCT02973984
Title: Evaluating the Efficacy and Risks of Anticoagulant Treatments in Multimorbid Frail Older Subjects With Atrial Fibrillation. The European Registry of Older Subjects With Atrial Fibrillation (EUROSAF)
Brief Title: The European Registry of Older Subjects With Atrial Fibrillation (EUROSAF)
Acronym: EUROSAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alberto Pilotto (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Alberto Pilotto, Director of Department Geriatric Care, OrthoGeriatrics and Rehabilitation, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Other Study IDs: 28UCS2015; 162REG2016 (Other: Ethics Commitee of the Liguria Region)
Record Dates: First submitted 2016-10-24; First posted 2016-11-28 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation
Keywords: Anticoagulant Treatments; Multidimensional Prognostic Index (MPI); Comprehensive Geriatric Assessment (CGA); Frailty; Elderly; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Preliminary data suggest that:

1. a different risk of mortality, as assessed by the Multidimensional Prognostic Indices (MPI), may influence the anticoagulant prescription in older subjects with Atrial Fibrillation (AF);
2. the presence of multidimensional impairment, disability and multi-morbidities are usually not included in the decision algorithm of the more appropriate treatments in older patients with AF;
3. considering the prognostic information, as calculated by the MPI, can be useful to physicians in identifying older patients with AF that can benefit from anticoagulant treatment in term of increased survival.

DETAILED DESCRIPTION:
The main objective of this observational study is to evaluate in a "real world" population of older hospitalized patients with AF, the clinical benefit/risk ratio of the anticoagulant treatments in terms of:

1. mortality (all-cause and vascular mortality);
2. thromboembolic events, i.e. stroke, systemic embolism;
3. bleeding side-effects, especially intracranial and gastrointestinal bleeding Secondary objective of the study is to evaluate whether a different prognostic profile, as determined by the MPI, is associated with 1) different kind of treatments for AF (no treatment vs anticoagulants, i.e. Vitamin K Antagonists (VKA) or novel oral anticoagulant (NOACs); and 2) differences in the main outcomes (i.e. mortality, major thromboembolic events and side effects including bleeding events).

ELIGIBILITY:
Inclusion Criteria:

This is an observational study in which all consecutive patients admitted to the Geriatrics Units involved in the project will be screened for inclusion. The inclusion criteria are:

1. patients of both genders, aged 65 years and older
2. admitted to hospital for acute diseases or a relapse of chronic diseases
3. with a documented diagnosis of non valvular AF
4. who are willing to participate in the survey and give their informed consent

Exclusion Criteria:

1. age less than 65 years
2. patients who have not provided informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This is a cross-national, prospective, observational study that will include about 3.000 older subjects (aged ≥ 65 years) with AF hospitalized in 30 European geriatric centers (about 100 subjects/center) for an acute disease or a relapse of a chronic diseases. The study is in the frame of the Special Interest Group on CGA (Comprehensive Geriatric Assessment) of the EUGMS (European Union Geriatric Medicine Society).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-11-18; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality and vascular mortality | 12 months
  Vascular mortality is defined as: stroke, embolism, myocardial infarction
thromboembolic events, | 12 months
  stroke and/or systemic embolism
bleeding side-effects | 12 months
  major intracranial and gastrointestinal bleeding.

SECONDARY OUTCOMES:
vascular-related hospitalization rates | 12 months
  stroke and/or systemic embolism
bleeding-related hospitalization rates | 12 months
  intracranial and gastrointestinal bleeding
MPI value and different mortality risk class | 12 months
  mild, moderate, severe
presence/absence of anticoagulant treatments | 12 months
  presence of anticoagulant treatments

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pilotto, MD, Principal Investigator — Dipartimento: area delle cure geriatriche, ortogeriatria e riabilitazione - E.O. Ospedali Galliera - Genova Italy
Locations (1):
- S.C. Geriatria, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Wann LS, Curtis AB, Ellenbogen KA, Estes NA 3rd, Ezekowitz MD, Jackman WM, January CT, Lowe JE, Page RL, Slotwiner DJ, Stevenson WG, Tracy CM, Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Le Heuzey JY, Kay GN, Olsson SB, Prystowsky EN, Tamargo JL, Wann S. Management of patients with atrial fibrillation (compilation of 2006 ACCF/AHA/ESC and 2011 ACCF/AHA/HRS recommendations): a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 May 7;61(18):1935-44. doi: 10.1016/j.jacc.2013.02.001. Epub 2013 Apr 1. No abstract available. PMID 23558044
- [Background] Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH; ESC Committee for Practice Guidelines. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Europace. 2010 Oct;12(10):1360-420. doi: 10.1093/europace/euq350. No abstract available. PMID 20876603
- [Background] Hylek EM, D'Antonio J, Evans-Molina C, Shea C, Henault LE, Regan S. Translating the results of randomized trials into clinical practice: the challenge of warfarin candidacy among hospitalized elderly patients with atrial fibrillation. Stroke. 2006 Apr;37(4):1075-80. doi: 10.1161/01.STR.0000209239.71702.ce. Epub 2006 Mar 9. PMID 16527999
- [Background] Pugh D, Pugh J, Mead GE. Attitudes of physicians regarding anticoagulation for atrial fibrillation: a systematic review. Age Ageing. 2011 Nov;40(6):675-83. doi: 10.1093/ageing/afr097. Epub 2011 Aug 5. PMID 21821732
- [Background] Maes F, Dalleur O, Henrard S, Wouters D, Scavee C, Spinewine A, Boland B. Risk scores and geriatric profile: can they really help us in anticoagulation decision making among older patients suffering from atrial fibrillation? Clin Interv Aging. 2014 Jul 15;9:1091-9. doi: 10.2147/CIA.S62597. eCollection 2014. PMID 25053883
- [Background] Sinnaeve PR, Brueckmann M, Clemens A, Oldgren J, Eikelboom J, Healey JS. Stroke prevention in elderly patients with atrial fibrillation: challenges for anticoagulation. J Intern Med. 2012 Jan;271(1):15-24. doi: 10.1111/j.1365-2796.2011.02464.x. Epub 2011 Oct 31. PMID 21995885
- [Background] Zarraga IG, Kron J. Oral anticoagulation in elderly adults with atrial fibrillation: integrating new options with old concepts. J Am Geriatr Soc. 2013 Jan;61(1):143-50. doi: 10.1111/jgs.12042. Epub 2012 Dec 18. PMID 23252345
- [Background] Barco S, Cheung YW, Eikelboom JW, Coppens M. New oral anticoagulants in elderly patients. Best Pract Res Clin Haematol. 2013 Jun;26(2):215-24. doi: 10.1016/j.beha.2013.07.011. Epub 2013 Jul 21. PMID 23953909
- [Background] Sardar P, Chatterjee S, Chaudhari S, Lip GY. New oral anticoagulants in elderly adults: evidence from a meta-analysis of randomized trials. J Am Geriatr Soc. 2014 May;62(5):857-64. doi: 10.1111/jgs.12799. Epub 2014 May 1. PMID 24786913
- [Background] Stollberger C, Finsterer J. Concerns about the use of new oral anticoagulants for stroke prevention in elderly patients with atrial fibrillation. Drugs Aging. 2013 Dec;30(12):949-58. doi: 10.1007/s40266-013-0119-3. PMID 24170233
- [Background] Crome P, Lally F, Cherubini A, Oristrell J, Beswick AD, Clarfield AM, Hertogh C, Lesauskaite V, Prada GI, Szczerbinska K, Topinkova E, Sinclair-Cohen J, Edbrooke D, Mills G. Exclusion of older people from clinical trials: professional views from nine European countries participating in the PREDICT study. Drugs Aging. 2011 Aug 1;28(8):667-77. doi: 10.2165/11591990-000000000-00000. PMID 21812501
- [Background] Gill TM. The central role of prognosis in clinical decision making. JAMA. 2012 Jan 11;307(2):199-200. doi: 10.1001/jama.2011.1992. No abstract available. PMID 22235093
- [Background] Pilotto A, Ferrucci L, Franceschi M, D'Ambrosio LP, Scarcelli C, Cascavilla L, Paris F, Placentino G, Seripa D, Dallapiccola B, Leandro G. Development and validation of a multidimensional prognostic index for one-year mortality from comprehensive geriatric assessment in hospitalized older patients. Rejuvenation Res. 2008 Feb;11(1):151-61. doi: 10.1089/rej.2007.0569. PMID 18173367
- [Background] Pilotto A, Gallina P, Fontana A, Sancarlo D, Bazzano S, Copetti M, Maggi S, Paroni G, Marcato F, Pellegrini F, Donato D, Ferrucci L. Development and validation of a Multidimensional Prognostic Index for mortality based on a standardized Multidimensional Assessment Schedule (MPI-SVaMA) in community-dwelling older subjects. J Am Med Dir Assoc. 2013 Apr;14(4):287-92. doi: 10.1016/j.jamda.2013.01.005. Epub 2013 Feb 9. PMID 23402948
- [Background] Siontis GC, Tzoulaki I, Ioannidis JP. Predicting death: an empirical evaluation of predictive tools for mortality. Arch Intern Med. 2011 Oct 24;171(19):1721-6. doi: 10.1001/archinternmed.2011.334. Epub 2011 Jul 25. PMID 21788535
- [Background] Yourman LC, Lee SJ, Schonberg MA, Widera EW, Smith AK. Prognostic indices for older adults: a systematic review. JAMA. 2012 Jan 11;307(2):182-92. doi: 10.1001/jama.2011.1966. PMID 22235089
- [Background] Pilotto A, Rengo F, Marchionni N, Sancarlo D, Fontana A, Panza F, Ferrucci L; FIRI-SIGG Study Group. Comparing the prognostic accuracy for all-cause mortality of frailty instruments: a multicentre 1-year follow-up in hospitalized older patients. PLoS One. 2012;7(1):e29090. doi: 10.1371/journal.pone.0029090. Epub 2012 Jan 11. PMID 22247767
- [Background] Volpato S, Bazzano S, Fontana A, Ferrucci L, Pilotto A; MPI-TriVeneto Study Group. Multidimensional Prognostic Index predicts mortality and length of stay during hospitalization in the older patients: a multicenter prospective study. J Gerontol A Biol Sci Med Sci. 2015 Mar;70(3):325-31. doi: 10.1093/gerona/glu167. Epub 2014 Sep 9. PMID 25209253
- [Background] Pilotto A, Panza F, Ferrucci L. A multidimensional prognostic index in common conditions leading to death in older patients. Arch Intern Med. 2012 Apr 9;172(7):594; discussion 594-5. doi: 10.1001/archinternmed.2011.1891. No abstract available. PMID 22493470
- [Background] Angleman SB, Santoni G, Pilotto A, Fratiglioni L, Welmer AK; MPI_AGE Project Investigators. Multidimensional Prognostic Index in Association with Future Mortality and Number of Hospital Days in a Population-Based Sample of Older Adults: Results of the EU Funded MPI_AGE Project. PLoS One. 2015 Jul 29;10(7):e0133789. doi: 10.1371/journal.pone.0133789. eCollection 2015. PMID 26222546
- [Background] Cerreta F, Eichler HG, Rasi G. Drug policy for an aging population--the European Medicines Agency's geriatric medicines strategy. N Engl J Med. 2012 Nov 22;367(21):1972-4. doi: 10.1056/NEJMp1209034. No abstract available. PMID 23171092
- [Background] Granziera S, Cohen AT, Nante G, Manzato E, Sergi G. Thromboembolic prevention in frail elderly patients with atrial fibrillation: a practical algorithm. J Am Med Dir Assoc. 2015 May 1;16(5):358-64. doi: 10.1016/j.jamda.2014.12.008. Epub 2015 Feb 11. PMID 25680239
- [Background] Olesen JB, Lip GY, Hansen ML, Hansen PR, Tolstrup JS, Lindhardsen J, Selmer C, Ahlehoff O, Olsen AM, Gislason GH, Torp-Pedersen C. Validation of risk stratification schemes for predicting stroke and thromboembolism in patients with atrial fibrillation: nationwide cohort study. BMJ. 2011 Jan 31;342:d124. doi: 10.1136/bmj.d124. PMID 21282258
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Derived] Pilotto A, Veronese N, Polidori MC, Strandberg T, Topinkova E, Cruz-Jentoft AJ, Custodero C, Maggi S; EUROSAF Study Investigators. The role of prognostic stratification on prescription of anticoagulants in older patients with atrial fibrillation: a multicenter, observational, prospective European study (EUROSAF). Ann Med. 2022 Dec;54(1):2411-2419. doi: 10.1080/07853890.2022.2117407. PMID 36062815
- [Derived] Veronese N, Argusti A, Canepa E, Polidori MC, Maggi S, Strandberg T, Pilotto A; EUROSAF Study Investigators. Evaluating the effectiveness and risks of oral anticoagulant treatments in multimorbid frail older subjects with atrial fibrillation using the multidimensional prognostic index: the EURopean study of older subjects with atrial fibrillation-EUROSAF. Eur Geriatr Med. 2018 Apr;9(2):149-154. doi: 10.1007/s41999-018-0026-6. Epub 2018 Feb 27. PMID 34654263